CLINICAL TRIAL: NCT00182702
Title: A Phase II Trial of BMS 247550 (Ixabepilone) in Advanced Renal Cell Carcinoma
Brief Title: Ixabepilone in Treating Patients With Metastatic, Recurrent, or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02669; 13850A; N01CM62201 (NIH); N01CM62209 (NIH); CDR0000440071 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — ixabepilone

ARMS (1):
- Treatment (Experimental): Patients receive ixabepilone IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ixabepilone; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well ixabepilone works in treating patients with metastatic, recurrent, or unresectable kidney cancer. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with metastatic, recurrent, or unresectable renal cell carcinoma treated with ixabepilone.

SECONDARY OBJECTIVES:

I. Determine the progression-free and overall survival rates in patients treated with this drug.

II. Determine the toxicity of this drug in these patients. III. Correlate VHL gene mutations with response in patients treated with this drug.

IV. Correlate VHL pathway protein expression with response in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive ixabepilone IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 9 weeks until disease progression and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma of 1 of the following subtypes:

  * Clear cell
  * Papillary, type I or II
  * Chromophobe
  * Collecting duct
  * Medullary
* Metastatic, recurrent, or unresectable disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No known active brain metastases requiring steroid or anticonvulsant therapy

  * Patients with definitively treated brain metastases are eligible provided they are not on steroids or anticonvulsants AND show no evidence of disease progression for ≥ 3 months after completion of definitive therapy
* Performance status - ECOG 0-2
* At least 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Glomerular filtration rate ≥ 50 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No HIV positivity
* No peripheral neuropathy > grade 1
* No psychiatric illness or social situation that would preclude study compliance
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drug
* No history of severe hypersensitivity reaction to agents containing Cremophor® EL
* No other active malignancy

  * Curatively treated malignancies are allowed provided the risk of recurrent disease at the time of study enrollment is < 20%
* No other uncontrolled illness
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior tubule inhibitors, including, but not limited to, any of the following:

  * Vinca alkaloids (e.g., vinblastine, vincristine, or vinorelbine)
  * Taxanes (e.g., docetaxel or paclitaxel)
  * Epothilones
* No other concurrent chemotherapy
* See Disease Characteristics
* No concurrent hormonal therapy except steroids for adrenal failure or hypersensitivity prophylaxis or hormones for non-disease related conditions (e.g., insulin for diabetes)
* More than 4 weeks since prior radiotherapy and recovered
* No concurrent palliative radiotherapy
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-07; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (partial or complete) | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the start of treatment to time of progression, assessed up to 5 years
  PFS rate will be estimated using the Kaplan-Meier method. Median PFS time and its associated 90% confidence interval will be estimated using the method of Brookmeyer and Crowley.
Overall survival (OS) | Up to 5 years
  OS rate will be estimated using the Kaplan-Meier method. Median OS time and its associated 90% confidence interval will be estimated using the method of Brookmeyer and Crowley.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States